CLINICAL TRIAL: NCT05157568
Title: Rethinking Post-acute Cardiac Care: Pilot Randomized Clinical Trial of Live-streamed Cardiovascular Rehabilitation
Brief Title: Pilot Randomized Clinical Trial of Live-streamed Cardiovascular Rehabilitation
Acronym: VirtualEX
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20210752-01H
Record Dates: First submitted 2021-12-01; First posted 2021-12-15 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Cardiac Disease
Keywords: Cardiovascular Rehabilitation; Virtual Rehabilitation
MeSH Terms: conditions — Heart Diseases | interventions — Equipment and Supplies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (C) (Active Comparator): Participants will receive a exercise prescription and a home exercise plan. It will specify how many days per week they should exercise and will indicate how hard they should be working using their heart rate and rating of perceived exertion (RPE) as a guide. They will attend 8 onsite rehabilitation classes at the University of Ottawa Heart Institute (1 class per week for 8 weeks). These classes will be led by a specially trained instructor who will teach and encourage self-monitoring of heart rate and RPE. The class will include a warm-up, 30 minutes of aerobic exercise and a 15 min cool-down, including strength exercises and stretches. Following each class there will be a short mini-education session highlighting a variety of topics on how to manage risk factors. Patients will have access to onsite classes for nutrition and stress management. Participants will receive access to 8 additional educational videos that highlight topics such as exercise safety, goal setting and nutrition.
  Interventions: Behavioral: Control
- Exercise Streaming (ES) (Active Comparator): Participants will complete 1 "live" virtual class per week for 8-weeks. Classes will be led by a specially trained instructor and will include a warm-up, 30 minutes of aerobic exercise, 10 minutes of strength exercises, and a cooldown and stretching segment. During each live class, the instructor will play the corresponding video and supervise the participants through the Zoom for Healthcare platform. Heart rates and RPE data will be collected from each participant. Participants will have access to other pre-recorded exercise videos that they can stream "on demand" at any time. They will be encouraged to access them "on demand" throughout the week. In addition participants will have access to the same 8 pre-recorded educational videos that the control group will receive. Topics include; exercise safety, goal setting, nutrition, stress management, medication information, risk factor awareness and transition planning.
  Interventions: Behavioral: Exercise Streaming (ES)
- Exercise Streaming + Equipment (ES+E) (Active Comparator): Participants will receive an indoor bicycle and an exercise band (delivered and set up in their home). Participants will complete 1 "live" class per week for 8 weeks. Their exercise prescription will be based on a stress test. Classes will be led by a specially trained instructor and will include a warm-up, 30 minutes of aerobic exercise, 10 minutes of strength exercises, and a cooldown and stretching segment. During each "live" class, the exercise supervisor will play the corresponding video and supervise the participants through the Zoom for Healthcare platform. Heart rate and RPE data will be collected from each participant. Participants will have access to other pre-recorded exercise videos that they can stream "on demand" at any time. Participants will be encouraged to access them throughout the week. Participants will have access to the same 8 pre-recorded educational videos that the control and exercise streaming groups will receive.
  Interventions: Behavioral: Exercise Streaming + Equipment (ES+E)

INTERVENTIONS:
Behavioral: Exercise Streaming (ES) — Participants will complete 8 weeks (1 class per week) of supervised exercise online. No equipment is required. They will follow a pre-recorded exercise video and at the same time, get instruction, feedback and support from their coach. Each class will be held as a teleconference.
  Arms: Exercise Streaming (ES)
Behavioral: Exercise Streaming + Equipment (ES+E) — Participants will complete 8 weeks (1 class per week) of supervised exercise online. Each participant will have a stationary exercise bike delivered to their home for use during their live classes. They will follow a pre-recorded exercise video and at the same time, get instruction, feedback and support from their coach. Each class will be held as a teleconference.
  Arms: Exercise Streaming + Equipment (ES+E)
Behavioral: Control — Participants will complete 8 weeks (1 class per week) of in-person supervised exercise.
  Arms: Control (C)

SUMMARY:
Cardiovascular Rehabilitation (CR) programs are designed to help people recover following a heart attack, heart surgery, or diagnosis of heart disease. Counseling, education, risk factor management, and efforts to increase levels of MVPA constitute the largest components of CR programs. Technological advances in video-conferencing and video-streaming are affording new opportunities to increase access to CR services and supervised exercise sessions for patients who are social distancing, or who face access issues (e.g., time, mobility, transportation etc.). Comfort with these technologies for CR staff and patients has been accelerated by the current pandemic. Technology-enabled interactions between patients and providers is a significant opportunity to help mitigate these effects. We developed a new model for delivery of group exercise training for people with heart disease. Our model delivers all the core components of CR (i.e. counseling, education, risk factor management) but also includes live-streaming of CR exercise classes. Two versions of these classes are available: one that does not require any exercise equipment; and one that relies on a stationary exercise bike and exercise band delivered and installed in patients' homes. The new model has performed well in proof-of-concept testing, but now needs to be rigorously evaluated.

DETAILED DESCRIPTION:
Heart diseases affect an estimated 2 million Canadians each year; they are chronic conditions that require patients to manage their health on a daily basis. Moderate-to-vigorous intensity aerobic exercise (e.g. walking, running, cycling) is a key self-management strategy for people living with heart disease and those who accumulate at least 150 minutes of moderate-to-vigorous intensity physical activity (MVPA) each week improve critical patient-relevant outcomes like cardiorespiratory fitness, symptoms of anxiety and depression, quality of life, rehospitalization, and mortality.

Cardiovascular Rehabilitation (CR) programs are designed to help people recover following a heart attack, heart surgery, or diagnosis of heart disease. Counseling, education, risk factor management, and efforts to increase levels of MVPA constitute the largest components of CR programs. In Canada, many patients with heart disease do not access CR programs. Estimates of the proportion of patients with heart disease that attend CR range from 22-52% and a majority of them are men. Long travel distance to CR centres, severe weather, work and caregiving responsibilities, other time constraints, and the costs for parking while attending CR programs consistently top patient-related barriers to participation. In addition, the current COVID-19 pandemic has forced CR programs to limit participation in on-site activities, significantly impacting the ability to provide exercise testing and supervised exercise training sessions, therapies known to improve outcomes. Many CR programs have switched to virtual care, a case-managed approach that is delivered by phone, email and/or the Internet. Participant feedback indicates drawbacks to home-based programming, including: a lack of social support (compared to on-site group exercise); a lack of instruction and feedback on exercise performance; a lack of appropriate home exercise equipment; and, a lack of structure for completing daily exercise sessions.

Technological advances in video-conferencing and video-streaming are affording new opportunities to increase access to CR services and supervised exercise sessions for patients who are social distancing, or who face access issues (e.g., time, mobility, transportation etc.). Comfort with these technologies for CR staff and patients has been accelerated by the current pandemic. Current and future pandemics are likely to feature waves of infection necessitating frequent and long periods of physical distancing, isolation, and healthcare disruption, particularly for vulnerable populations, such as those with heart disease. This will result in progressively poorer physical and mental health for people living with these conditions. Technology-enabled interactions between patients and providers is a significant opportunity to help mitigate these effects.

Few randomized controlled trials (RCT) of real-time, video-conferencing-based exercise rehabilitation have been conducted. A scoping review of digital cardiology applications did not include any video-conference-based supervised exercise interventions. We conducted literature searches using the terms 'video-conference,' 'randomized trial,' and 'exercise' and identified only 2 published studies. Tsai and colleagues randomized 37 patients with COPD to either a supervised, home-based tele-rehabilitation group that received exercise training via videoconference 3 times/week for 8 weeks, or a control group that received usual care without exercise training. After 8 weeks, participants in the intervention group showed a significant increase in endurance shuttle walk test time compared to participants in the control group (between group difference = 340 s; P <.0001) (7). Duruturk and Oskoslu randomized 50 participants with type 2 diabetes to treatment or control. Participants in the treatment group performed breathing and calisthenic exercises, three times a week, for 6 weeks, at home by Internet-based video conferences. HbA1c (P <.01), 6 min walking distance (P <.01), and depression levels (P <.01) changed significantly in the treatment versus the control group.

The incremental value of installing specific forms of home exercise equipment is also an important question. Proper equipment may allow people to increase the volume and intensity of their workouts, important drivers of adaptation to exercise and improvements in cardiorespiratory and functional fitness. We were able to locate only one RCT in patients with chronic illness that used provision of home exercise equipment as an independent variable. Jakicic et al examined the effects of home exercise equipment in 148 overweight women (9). Participants who had a treadmill installed in their home achieved greater weight loss (-7.4 kg vs. -3.7 kg; P <.05) and completed more exercise sessions each week in follow-up compared to participants receiving exercise coaching only (6.6 vs. 4.3 sessions per week; P <.05). Of note, the pandemic has accelerated adoption of home exercise equipment and exercise class streaming among healthy adults (e.g. Peloton, Mirror); none of these applications are designed to meet the needs of people with heart disease.

We developed a new model for delivery of group exercise training for people with heart disease. Our model delivers all the core components of CR (i.e. counseling, education, risk factor management) but also includes live-streaming of CR exercise classes. Two versions of these classes are available: one that does not require any exercise equipment; and one that relies on a stationary exercise bike and exercise band delivered and installed in patients' homes. The new model has performed well in proof-of-concept testing, but now needs to be rigorously evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Patient was discharged from hospitalized at UOHI within the last 12 weeks;
2. Patient has stable CHD or repaired valvular disease;
3. Patient has been referred to CR and is a candidate an offsite program;
4. Patient is able to completed a cardiopulmonary exercise test;
5. Patient has access to and regularly uses a smart phone, tablet or computer with Internet access;
6. Patient is ≥ 18 years of age (the age of consent in Ontario);
7. Patient is able to provide informed consent

Exclusion Criteria:

1. Patient was hospitalized for heart failure, congenital heart disease, transplant or arrhythmia within the last 6 months;
2. Patient, in the opinion of the medical advisor (Dr. Andrew Pipe/Dr. Hassan Mir), manifests illness or disease that would preclude participation in the interventions (e.g. cognitive impairment, active drug or alcohol dependence, unresolved cardiac symptoms).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-09-20 (Actual); Primary Completion 2023-02-24 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Eligibility | 8 weeks
  What proportion of patients referred to CR are eligible to participate based on the inclusion and exclusion criteria?
Feasibility of recruitment | 8 weeks
  What proportion of eligible patients accept the invitation to participate in the research and agree to be randomized to treatment?
Feasibility of equipment delivery | 8 weeks
  Are the interventions acceptable in terms of completion of delivery and set-up of home exercise equipment (ES+E group only), scheduled coaching contacts, and exercise training class attendance (ES and ES+E groups)?
Retention | 8 weeks
  How many patients will complete of follow-up assessments at the end of intervention (8 weeks)?

CONTACTS AND LOCATIONS:
Overall Officials: Thais Coutinho, MD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- The University of Ottawa Heart Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No